CLINICAL TRIAL: NCT01220999
Title: A Phase I Imaging and Pharmacodynamic Trial of CS-1008 in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUD2010-002
Record Dates: First submitted 2010-10-12; First posted 2010-10-14 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Neoplasms
Keywords: Clinical trial; CS-1008 mAb; monoclonal antibody CS-1008; Positron-Emission Tomography; Pharmacokinetics; Pharmacodynamics; apoptosis; caspases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tigatuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Subjects received an initial loading dose of 111^In-CS-1008 (0.2 mg/kg) on Day 1, CS-1008 (6 mg/kg) on Day 8, and subsequent weekly doses of CS-1008 (2 mg/kg) on Days 15, 22, 29, 36, and 43; the Day 36 dose was also radiolabeled with 111^In. Additional 4-week cycles of weekly CS-1008 (2 mg/kg) were permitted for subjects benefiting from treatment.
  Interventions: Drug: CS-1008
- Cohort 2 (Experimental): Subjects received an initial loading dose of 111^In-CS-1008 (1 mg/kg) on Day 1, CS-1008 (6 mg/kg) on Day 8, and subsequent weekly doses of CS-1008 (2 mg/kg) on Days 15, 22, 29, 36, and 43; the Day 36 dose was also radiolabeled with 111^In. Additional 4-week cycles of weekly CS-1008 (2 mg/kg) were permitted for subjects benefiting from treatment.
  Interventions: Drug: CS-1008
- Cohort 3 (Experimental): Subjects received an initial loading dose of 111^In-CS-1008 (2 mg/kg) on Day 1, CS-1008 (6 mg/kg) on Day 8, and subsequent weekly doses of CS-1008 (2 mg/kg) on Days 15, 22, 29, 36, and 43; the Day 36 dose was also radiolabeled with 111^In. Additional 4-week cycles of weekly CS-1008 (2 mg/kg) were permitted for subjects benefiting from treatment.
  Interventions: Drug: CS-1008
- Cohort 4 (Experimental): Subjects received an initial loading dose of 111^In-CS-1008 (4 mg/kg) on Day 1, CS-1008 (4 mg/kg) on Day 8, and subsequent weekly doses of CS-1008 (2 mg/kg) on Days 15, 22, 29, 36, and 43; the Day 36 dose was also radiolabeled with 111^In. Additional 4-week cycles of weekly CS-1008 (2 mg/kg) were permitted for subjects benefiting from treatment.
  Interventions: Drug: CS-1008
- Cohort 5 (Experimental): Subjects received an initial loading dose of 111^In-CS-1008 (6 mg/kg) on Day 1, CS-1008 (2 mg/kg) on Day 8, and subsequent weekly doses of CS-1008 (2 mg/kg) on Days 15, 22, 29, 36, and 43; the Day 36 dose was also radiolabeled with 111^In. Additional 4-week cycles of weekly CS-1008 (2 mg/kg) were permitted for subjects benefiting from treatment.
  Interventions: Drug: CS-1008

INTERVENTIONS:
Drug: CS-1008 — CS-1008 was administered once weekly as an intravenous infusion over 30 ± 10 minutes at a dose range of 0.2 to 6 mg/kg. On Days 1 and 36, CS-1008 infusions were radiolabeled with 111^In (5-7 mCi).
  Other Names: Tigatuzumab

SUMMARY:
This was a Phase 1, open-label, single-center study of CS-1008, an immunoglobulin G subclass 1 (IgG1) humanized monoclonal antibody, in subjects with advanced colorectal carcinoma who had received ≥ 1 prior chemotherapy regimen for metastatic disease. Primary study objectives were to determine the influence of the CS-1008 dose on the biodistribution, pharmacokinetics (PK) and tumor uptake of radiolabeled CS-1008 following a single infusion and following continuous sequential doses of CS-1008. Secondary objectives were to evaluate changes in tumor metabolism, antitumor response, and changes in serum apoptosis biomarkers and tumor response markers following treatment with CS-1008.

DETAILED DESCRIPTION:
Eligible subjects were to be enrolled into one of 5 dose-escalation cohorts to receive CS-1008 administered weekly as an intravenous (IV) infusion over 30 ± 10 minutes. Each cohort initially comprised 2 subjects but was expanded in up to 5 subjects if additional biodistribution and/or PK data were required.

The initial infusion of CS-1008 on Day 1 was trace labeled with Indium-111 (111^In-CS-1008; 5-7 mCi) and was investigated at escalating doses up to the standard loading dose, as follows: Cohort 1 (0.2 mg/kg), Cohort 2 (1 mg/kg), Cohort 3 (2 mg/kg), Cohort 4 (4 mg/kg), and Cohort 5 (6 mg/kg). The initial 111^In-CS-1008 dose was followed by gamma camera imaging with blood sampling over a 10-day period to evaluate biodistribution, tumor uptake, PK, and serum biomarkers. Day 8 dosing comprised non-labeled CS-1008 at doses of 6 mg/kg in Cohorts 1-3, 4 mg/kg in Cohort 4, and 2 mg/kg in Cohort 5. Subsequent weekly infusions of standard dose CS-1008 (2 mg/kg) were administered on Days 15, 22, 29, 36, and 43. The Day 36 infusion of CS-1008 was also trace labeled with 111^In (5-7 mCi), with subsequent gamma camera imaging and blood sampling.

Subjects were assessed for disease status using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, serum tumor biomarkers (carcinoembryonic antigen [CEA]), and human-anti-CS-1008-antibody development (HAHA). Subjects were assessed for changes in tumor metabolism following CS-1008 administration using computed tomography (CT) or fluorodeoxyglucose positron emission tomography (18^F-FDG PET) scans.

Cycle 1 encompassed the first 7 weeks of therapy. Within 1 week (Days 44-50) after the last infusion of CS-1008, subjects completed an End of Study/End of Cycle 1 assessment. Subjects with stable disease or better (according to RECIST version 1.1) at the Day 44-50 reassessment were permitted to receive additional 4-week cycles of CS-1008 (2 mg/kg) until disease progression, unacceptable toxicity, or subject/physician decision.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven metastatic colorectal cancer with 1 target lesion ≥ 2 cm and evaluable by gamma camera imaging. If this lesion was previously irradiated, progression must have been documented following radiotherapy.
2. Received at least 1 prior course of chemotherapy for metastatic disease.
3. Expected survival of at least 3 months.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
5. Age ≥ 18 years old.
6. Able and willing to give valid written informed consent.
7. Within the last 1 week prior to first study drug administration, laboratory parameters for vital functions were to be in the normal range. Laboratory abnormalities that were not clinically significant were generally permitted, except for the following laboratory parameters, which were to be within the ranges specified:

   * Neutrophil count: ≥ 1.5 x 10^9/L
   * Platelet count: ≥ 90 x 10^9/L
   * International normalized ratio: ≤ 1.5
   * Serum bilirubin: ≤ 1.5 x upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT): ≤ 2 x ULN (≤ 5 x ULN if liver metastases)
   * Calculated creatinine clearance (Cockcroft-Gault formula): ≥ 55 mL/min

Exclusion Criteria:

1. Active central nervous system metastases. Definitively treated metastases were allowed if stable for 6 weeks off therapy.
2. Known immunodeficiency or human immunodeficiency virus positivity.
3. Serious illnesses, e.g., serious infections requiring antibiotics, bleeding disorders, or any condition that in the opinion of the Investigator would have interfered with the ability of the subject to fulfill the study requirements.
4. Other malignancy, apart from non-melanoma skin cancer, within 3 years prior to first study drug administration, that in the opinion of the Investigator had >10% risk of relapse within 12 months.
5. Chemotherapy, radiotherapy, or investigational agent within 4 weeks prior to first study drug administration.
6. Regular corticosteroid, nonsteroidal anti-inflammatory drug (NSAID) (other than paracetamol or low-dose aspirin) or other immunosuppressive treatment within 3 weeks prior to first drug administration. Intermittent dosing of corticosteroid or NSAID was permitted if less than 4 doses within a 3-day period.
7. Mental impairment that may have compromised the ability to give informed consent and comply with the requirements of the study.
8. Lack of availability for clinical follow-up assessments.
9. Pregnancy or breastfeeding.
10. Women of childbearing potential: refusal or inability to use effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-10-12 (Actual); Primary Completion 2012-06-27 (Actual); Study Completion 2012-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Scott, MBBS, MD, FRACP, DDU, Principal Investigator — Ludwig Institute for Cancer Research & Austin Health
Locations (1):
- Ludwig Institute Tumor Targeting Program, Austin Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Young H, Baum R, Cremerius U, Herholz K, Hoekstra O, Lammertsma AA, Pruim J, Price P. Measurement of clinical and subclinical tumour response using [18F]-fluorodeoxyglucose and positron emission tomography: review and 1999 EORTC recommendations. European Organization for Research and Treatment of Cancer (EORTC) PET Study Group. Eur J Cancer. 1999 Dec;35(13):1773-82. doi: 10.1016/s0959-8049(99)00229-4. PMID 10673991
- [Result] Ciprotti M, Tebbutt NC, Lee FT, Lee ST, Gan HK, McKee DC, O'Keefe GJ, Gong SJ, Chong G, Hopkins W, Chappell B, Scott FE, Brechbiel MW, Tse AN, Jansen M, Matsumura M, Kotsuma M, Watanabe R, Venhaus R, Beckman RA, Greenberg J, Scott AM. Phase I Imaging and Pharmacodynamic Trial of CS-1008 in Patients With Metastatic Colorectal Cancer. J Clin Oncol. 2015 Aug 20;33(24):2609-16. doi: 10.1200/JCO.2014.60.4256. Epub 2015 Jun 29. PMID 26124477
- See also: Full-text of Ciprotti et al 2015 — http://ascopubs.org/doi/pdf/10.1200/JCO.2014.60.4256

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 2 | 4 | 5 | 3 | 5
Completed (Completed Cycle 1 (through Day 43) as planned) | 2 | 4 | 4 | 3 | 5
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 2 | 4 | 5 | 3 | 5 | 19
Age, Continuous [Median (Full Range); unit: years] | 66.0 [64 to 68] | 60.5 [52 to 65] | 65.0 [50 to 74] | 65.0 [57 to 83] | 63.0 [51 to 80] | 64.0 [50 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 2 | 2 | 8
  Male | 2 | 2 | 3 | 1 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 4 | 5 | 3 | 5 | 19
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 2 | 4 | 5 | 3 | 5 | 19
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Median (Full Range); unit: units on a scale] — PS 0 = Fully active, able to carry on all pre-disease performance without restriction; PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; PS 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; PS 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; PS 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; PS 5 = Dead
  units on a scale | 0.5 [0 to 1] | 0.0 [0 to 1] | 1.0 [0 to 1] | 1.0 [1 to 1] | 1.0 [0 to 2] | 1.0 [0 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Tumor Uptake of 111^In-CS-1008 in Target Lesions Based on Gamma Camera Imaging Following the Day 1 and Day 36 Infusions
Description: Tumor localization was assessed using gamma camera imaging performed after the initial infusion of 111^In-CS-1008 on Day 1 and then on Days 2, 4/5, 7/8, and 11/12 (collectively, "After Day 1 Infusion" in the table) and after the second infusion of 111^In-CS-1008 on Day 36 and then on Days 37, 39/40, and 42/43 (collectively, "After Day 36 Infusion" in the table). Dosimetry calculations were performed to determine the tumor localization properties of 111^In-CS-1008. Calculation of whole body dose and doses to individual organs by 111^In-CS-1008 were performed based on conjugate view images obtained from quantitative whole body images obtained at multiple time points. MIRD formalism was used in the calculation of doses.
Time Frame: Up to 43 days
Population: The population comprises all subjects who completed study requirements through Cycle 1 (Day 43). One patient in Cohort 3 was prematurely withdrawn from the study on Day 36 due to symptomatic deterioration secondary to progressive disease (radiologically documented) and did not complete Cycle 1.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 2 | 4 | 5 | 3 | 5
participants
  After Day 1 infusion: High, Specific Uptake | 0 | 3 | 3 | 3 | 3
  After Day 1 infusion: No Uptake | 2 | 1 | 2 | 0 | 2
  After Day 36 infusion: High, Specific Uptake: number analyzed (Participants) | 2 | 4 | 4 | 3 | 5
  After Day 36 infusion: High, Specific Uptake | 0 | 3 | 3 | 3 | 3
  After Day 36 infusion: No Uptake: number analyzed (Participants) | 2 | 4 | 4 | 3 | 5
  After Day 36 infusion: No Uptake | 2 | 1 | 1 | 0 | 2

2. Primary Outcome: Mean Tumor Uptake of 111^In-CS-1008 Based on Gamma Camera Imaging Following the Day 1 and Day 36 Infusions
Description: Tumor localization was assessed using gamma camera imaging performed on Days 7/8 and 42/43. Dosimetry calculations were performed to determine the tumor localization properties of 111^In-CS-1008. Calculation of whole body dose and doses to individual organs by 111^In-CS-1008 were performed based on conjugate view images obtained from quantitative whole body images obtained at multiple time points. MIRD formalism was used in the calculation of doses.
Time Frame: Up to 43 days
Population: The population comprises all subjects who completed study requirements through Cycle 1 (Day 43) and had tumor uptake.
Measure: Mean (Standard Deviation); unit: % of injected dose/g of organ
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 3
% of injected dose/g of organ
  Post-infusion tumor uptake: Day 7/8 |  | 0.0042 (0.0013) | 0.0063 (0.0004) | 0.0044 (0.0015) | 0.0043 (0.0006)
  Post-infusion tumor uptake: Day 42/43 |  | 0.0045 (0.0005) | 0.0061 (0.0011) | 0.0044 (0.0012) | 0.0036 (0.0007)

3. Primary Outcome: Mean 111^In-CS-1008 Serum Half-life by Gamma Counting Following the Day 1 Infusion of 111^In-CS-1008
Description: The serum PK of CS-1008 was evaluated by gamma scintillation counting to assess serum radioactivity (111^In-CS-1008) and CS-1008 protein concentration following the Day 1 infusion at the following time points: Day 1 (pre-infusion and 5 minutes and 1, 2, and 4 hours post-infusion), Day 2 (24 hours after Day 1 infusion), Day 4/5, Day 7/8 (pre-infusion and 5 minutes post-infusion if on Day 8), Day 11/12, and Day 36 (pre-infusion).
Time Frame: Up to 36 days
Population: The population comprises all subjects who received Day 1 of study treatment and had post-infusion PK samples evaluable by gamma scintillation counting.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 2 | 4 | 5 | 2 | 4
hours
  Initial half-life | 14.51 (5.95) | 21.52 (5.76) | 5.29 (4.76) | 10.45 (6.85) | 14.73 (4.72)
  Terminal half-life | 284.76 (0.38) | 264.89 (122.12) | 163.08 (39.86) | 243.39 (52.21) | 247.5 (52.9)

4. Primary Outcome: Mean 111^In-CS-1008 Serum Volume of Central Compartment by Gamma Counting Following the Day 1 Infusion of 111^In-CS-1008
Description: as for outcome 3
Time Frame: Up to 36 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 2 | 4 | 5 | 2 | 4
mL | 3209.83 (321.96) | 2592.36 (303.21) | 3329.11 (624.49) | 2658.70 (112.60) | 4037 (425)

5. Primary Outcome: Mean 111^In-CS-1008 Serum Area Under the Curve by Gamma Counting Following the Day 1 Infusion of 111^In-CS-1008
Description: as for outcome 3
Time Frame: Up to 36 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*μg/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 2 | 4 | 5 | 2 | 4
hr*μg/mL | 986.58 (125.11) | 5706.38 (2632.72) | 8386.68 (855.70) | 18714.05 (1511.25) | 28492 (1598)

6. Primary Outcome: Mean 111^In-CS-1008 Serum Total Clearance by Gamma Counting Following the Day 1 Infusion of 111^In-CS-1008
Description: as for outcome 3
Time Frame: Up to 36 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 2 | 4 | 5 | 2 | 4
mL/hr | 14.92 (2.5) | 12.31 (3.38) | 18.23 (0.51) | 12 (2.03) | 18.52 (2.61)

7. Primary Outcome: Mean 111^In-CS-1008 Serum Maximum Concentration by Gamma Counting Following the Day 1 Infusion of 111^In-CS-1008
Description: as for outcome 3
Time Frame: Up to 36 days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 2 | 4 | 5 | 2 | 4
μg/mL | 4.59 (0.89) | 24.6 (3.75) | 47.29 (10.19) | 84.14 (11) | 131.3 (20.1)

8. Primary Outcome: Mean 111^In-CS-1008 Serum Half-life by Gamma Counting Following the Day 36 Infusion of 111^In-CS-1008
Description: The serum PK of CS-1008 was evaluated by gamma scintillation counting to assess serum radioactivity (111^In-CS-1008) and CS-1008 protein concentration following the Day 36 infusion at the following time points: Day 36 (pre-infusion and 5 minutes and 1, 2, and 4 hours post-infusion), Day 37 (24 hours after Day 36 infusion), Day 39/40, Day 43 (pre-infusion and 5 minutes post-infusion), and at the End of Cycle visit (Days 44-50).
Time Frame: Up to 50 days
Population: The population comprises all subjects who completed study requirements through Cycle 1 (Day 43) and had post-infusion PK samples evaluable by gamma scintillation counting.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 4 | 3 | 2 | 3
hours
  Initial half-life |  | 12.21 (6.13) | 15.84 (13.25) | 15.01 (3.48) | 15.56 (4.17)
  Terminal half-life |  | 186.2 (36.3) | 247.5 (109.3) | 347 (202) | 260.5 (51.1)

9. Primary Outcome: Mean 111^In-CS-1008 Serum Volume of Central Compartment by Gamma Counting Following the Day 36 Infusion of 111^In-CS-1008
Description: as for outcome 8
Time Frame: Up to 50 days
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 4 | 3 | 2 | 3
mL |  | 2510 (313) | 3272 (733) | 2742 (304) | 3985 (660)

10. Primary Outcome: Mean 111^In-CS-1008 Serum Area Under the Curve by Gamma Counting Following the Day 36 Infusion of 111^In-CS-1008
Description: as for outcome 8
Time Frame: Up to 50 days
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hr*μg/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 4 | 3 | 2 | 3
hr*μg/mL |  | 9013 (1629) | 9772 (626) | 10990 (3205) | 10465 (3286)

11. Primary Outcome: Mean 111^In-CS-1008 Serum Total Clearance by Gamma Counting Following the Day 36 Infusion of 111^In-CS-1008
Description: as for outcome 8
Time Frame: Up to 50 days
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 4 | 3 | 2 | 3
mL/hr |  | 14.11 (1.35) | 15.29 (2) | 10.73 (4.43) | 19.00 (6.48)

12. Primary Outcome: Mean 111^In-CS-1008 Serum Maximum Concentration by Gamma Counting Following the Day 36 Infusion of 111^In-CS-1008
Description: as for outcome 8
Time Frame: Up to 50 days
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 0 | 4 | 3 | 2 | 3
μg/mL |  | 51.08 (11.62) | 47.10 (12.07) | 40.98 (9.77) | 47.38 (9.99)

13. Secondary Outcome: Number of Subjects With Best Overall Tumor Response
Description: Tumor responses were evaluated using appropriate imaging and categorized according to the Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1, at Screening, at the end of every odd-numbered cycle (i.e., Cycles 1, 3, and 5, as applicable), and at the time of treatment discontinuation. Per RECIST 1.1, target lesions are categorized as follows: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria (Eisenhauer et al. Eur J Cancer 2009;45:228-47).
Time Frame: Up to 7 months
Population: The population comprises all subjects who received at least 1 dose of study treatment and had at least 1 applicable post-baseline response evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 2 | 4 | 5 | 3 | 5
Participants
  PR | 0 | 0 | 0 | 1 | 0
  SD | 1 | 2 | 2 | 2 | 1
  PD | 1 | 2 | 3 | 0 | 4

14. Secondary Outcome: Number of Subjects With Best Overall Metabolic Response
Description: Metabolic response to CS-1008 was assessed by fluorodeoxyglucose positron emission tomography (18^F-FDG PET) at Screening, Day 15, and at the End of Cycle 1/End of Study visit (Days 44-50). For each FDG-PET performed, the maximum standardized uptake value (SUVmax) corrected for body weight for all target lesions >2 cm identified on CT imaging was calculated using region of interest (ROI). The ROI was determined with the aid of the anatomical detail provided by the CT scan. Tumor metabolic response to CS-1008 was assessed by 18^F-FDG PET/CT calculated using the target lesion with the greatest baseline SUVmax, and was categorized according to the European Organization for Research and Treatment of Cancer (EORTC) guidelines (Young et al. Eur J Cancer 1999;35:1773-82).
Time Frame: Up to 50 days
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 2 | 4 | 5 | 3 | 5
Participants
  Metabolic PR | 0 | 0 | 0 | 1 | 0
  Metabolic SD | 1 | 2 | 3 | 2 | 0
  Metabolic PD | 1 | 2 | 2 | 0 | 5

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs that occurred or worsened in severity after the first dose of study treatment were considered treatment emergent (i.e., TEAEs). The AE reporting period for this study was up to 7 months.
Description: AE documentation included onset/resolution dates, severity using the NCI CTCAE (version 4.0), relationship to study drug, seriousness, study drug intervention, treatment, and outcome. In summaries, preferred terms were counted only once per subject at the maximum reported grade.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/5 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 3/5 | 1/3 | 0/5
Other Adverse Events (participants affected / at risk) | 2/2 | 2/4 | 3/5 | 3/3 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=2) | Cohort 2 (N=4) | Cohort 3 (N=5) | Cohort 4 (N=3) | Cohort 5 (N=5)
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=2) | Cohort 2 (N=4) | Cohort 3 (N=5) | Cohort 4 (N=3) | Cohort 5 (N=5)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes